CLINICAL TRIAL: NCT00324220
Title: A Phase I/II Study of MGCD0103 (MG-0103) in Combination With Azacitidine in Patients With High-Risk Myelodysplastic Syndrome or Acute Myelogenous Leukemia
Brief Title: A Phase I/II Study of MGCD0103 With Azacitidine in Patients With High-Risk Myelodysplastic Syndrome (MDS) or Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-005
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myelogenous Leukemia
Keywords: Phase I/II
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MGCD0103 oral administration 3 times per week.
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 Oral administration 3 times per week.

SUMMARY:
In this study, MGCD0103, a new anticancer drug under investigation, is given three times weekly in combination with azacitidine to patients with high-risk myelodysplastic syndromes or acute myelogenous leukemia.

DETAILED DESCRIPTION:
Phase I: The purpose of the first part (Phase 1) of this study is to find out what side effects the experimental drug MG-0103 in combination with azacitidine has on your body. The first part, or Phase, of the study will find out how much MG-0103 can be given safely along with azacitidine to people with cancer without causing side effects that are too severe. Patients are given MG-0103 and azacitidine and are watched closely to see what side effects may develop and to make sure that if side effects are seen, they can be taken care of rapidly. If the side effects are not severe, then more patients are asked to join the study and are given the same or a slightly higher dose of MG-0103. If there are no severe side effects, patients joining the study later on will get higher doses of MG-0103 than patients who join earlier. All patients will get the same dose of azacitidine. This will continue until a dose of MG-0103 is found that causes severe side effects in a high enough portion of patients. This will be the maximum dose of MG-0103 that can be given to patients in this study. Doses higher than that will not be given. Additional patients may be asked to join the study and receive MG-0103 and possibly azacitidine at lower doses that did not cause severe side effects.

Phase II: MG-0103 in combination with azacitidine may also have some effect on your disease. The purpose of the second part (Phase 2) of this study is to find out what, if any, effect there is. This Phase of the study will also find out more information about side effects of this combination of drugs. In this Phase, patients will receive a slightly lower dose than the maximum dose found in the first part of the study (which causes tolerable side effects). If a certain effect on the disease of patients is seen, then more patients are asked to join the study. Additional patients may also be asked to join the study and receive a lower dose if information collected during the study suggests that this should be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have high-risk MDS (≥ 10% BM blasts) or AML

  * RAEB (RA with excess blasts) with ≥10% BM blasts: 10%-20% blasts in BM, <5% blasts in peripheral blood
  * RAEB-T (RAEB in transformation): 21%-30% blasts in BM, <5% blasts in peripheral blood, absolute monocytosis (>109/L)
  * AML
* Disease may be relapsed/refractory or de novo. Once the MTD has been determined, all subsequent patients in the phase II portion of the study should have no prior azacitidine
* ECOG performance status of 0, 1, or 2
* Age ≥18 years
* Laboratory requirements
* Patients or their legal representative must be able to read, understand, and sign a written informed consent (approved by the institutional review board/Ethics Committee (IRB/EC)) within 14 days prior to start of treatment

Exclusion Criteria:

* Patients with another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia (CIN / cervical in situ)). Prior history of cancer is allowed, as long as there is no active disease
* Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test documented within 7 days prior start of study drug
* WOCBP and men whose partners are WOCBP must use an acceptable method of contraception while enrolled on this study, and for a period of 3 months following study drug treatment. Patients unwilling or unable to follow this guideline will be excluded. Examples of acceptable forms of contraception include an oral contraceptive or a double barrier method, such as condom with diaphragm
* Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever >38.5˚C on the day of scheduled dosing
* Patients with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
* Patients who have been treated with any investigational drug within 30 days prior to study initiation (an investigational drug is one for which there is no approved indication), or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy
* Known hypersensitivity to HDAC inhibitors, to any of the components of MG-0103 or Vidaza, including mannitol
* Prior treatment with azacitidine during the expanded phase II portion only
* Known HIV or active Hepatitis B or C
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and undergo study procedures
* Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures. For example, consider requirement to take MG-0103 with an acidic drink and recommendation to avoid agents that increase gastric-pH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose in combination with azacitidine | 1 year (anticipated)
Clinical response | 1 year (anticipated)

SECONDARY OUTCOMES:
Dose limiting toxicities | 1 year (anticipated)
Pharmacokinetics | 1 year (anticipated)
Objective response | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - St. Francis Hospital & Health Center, Beech Grove, Indiana
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas